CLINICAL TRIAL: NCT00740298
Title: Thermal Analgesia in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15480A; 5K23HD049452 (NIH)
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Pain
Keywords: infants; undergoing; vaccinations
MeSH Terms: conditions — Pain | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sweet Taste
  Interventions: Other: sucrose
- 2 (Active Comparator): warmth
  Interventions: Other: warmth

INTERVENTIONS:
Other: sucrose — sweet taste
  Arms: 1
Other: warmth — warmth
  Arms: 2

SUMMARY:
Newborns routinely experience pain associated with invasive procedures such as blood sampling, immunization, vitamin K injection, or circumcision. Prevention of pain is both an ethical expectation and a professional imperative, as untreated pain has deleterious consequences including altered pain sensitivity in later childhood and may be related to the permanent neuroanatomical and behavioral abnormalities as found in animal models. Moreover, pain is a source of concern and distress for new parents. Yet, pain reducing therapies are often underused for the numerous minor procedures that are a part of routine medical and nursing care for neonates. Growing scientific and clinical literature provides evidence for the effectiveness of natural, non-pharmacological techniques in both animal and human newborns. This study compares the pain reliving effects of sweet taste to the combination of sweet taste and warmth.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants

Exclusion Criteria:

* unhealthy infants

Max Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Decreased behavioral and physiologic indicators of pain | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Gray, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States